CLINICAL TRIAL: NCT06902857
Title: Prospective Observational Study on the Predictive Value of Cardiac Damage Markers High-sensitivity Cardiac Troponin I (Hs-cTnI), N-terminal Pro-B-natriuretic Peptide (NT-proBNP) and Soluble Suppression of Tumorigenesis-2 (sST2) for Mortality and the Development of Cardiovascular Events in Patients With Type 2 Diabetes (Diabetes-CV).
Brief Title: Study on the Predictive Value of High-sensitivity Cardiac Troponin I, N-terminal Pro-B-natriuretic Peptide, and Soluble Suppression of Tumorigenesis-2 for Mortality and the Development of Cardiovascular Events in Patients With Type 2 Diabetes (Diabetes-CV)
Acronym: Diabetes-CV
Status: Recruiting | Type: Observational
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Other Study IDs: INRCA_002_2025
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes; Cardiovascular Complication
Keywords: type 2 diabetes; high-sensitivity cardiac troponin I; N-terminal pro-B-natriuretic peptide; soluble suppression of tumorigenesis-2; mortality risk; diabetes complications
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma samples will be stored at -80°C at the BioGer biobank of IRCCS INRCA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with diabetes: Patients with type 2 diabetes attending routine check-ups at the Diabetology Unit outpatient clinic.

SUMMARY:
The Diabetes-CV study is an observational study designed to assess the prognostic value of serum cardiac damage markers high-sensitivity cardiac troponin I (hs-cTnI), N-terminal pro-B-natriuretic peptide (NT-proBNP), and soluble suppression of tumorigenesis-2 (sST2) in predicting mortality, major adverse cardiovascular events, and diabetic complications in patients with type 2 diabetes.

DETAILED DESCRIPTION:
This single-center, investigator-initiated, prospective observational study aims to evaluate the prognostic value of serum cardiac damage markers such as high-sensitivity cardiac troponin I (hs-cTnI), N-terminal pro-B-natriuretic peptide (NT-proBNP) and soluble suppression of tumorigenesis-2 (sST2) in subjects with type 2 diabetes. The study will utilize clinical and laboratory data from patients attending the Diabetology Unit at the IRCCS INRCA Hospital in Ancona (Italy), including both study-specific data and information extracted from routine outpatient medical records.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* patients attending the outpatient services

Exclusion Criteria:

* type 1 diabetes
* patients with active cancer or cancer in remission for less than 5 years
* any medical or other reason that leads the investigator to consider the subject ineligible for the study.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with type 2 diabetes attending the outpatient services for the routine checkups.
Sampling Method: Non-Probability Sample
Enrollment: 1002 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of all-cause mortality | From date of enrollment up to 36 months
  Death from any cause

SECONDARY OUTCOMES:
Change in high-sensitivity cardiac troponin I levels | At enrollment and 36 months later
  The levels of high-sensitivity cardiac troponin I will be analyzed.
The occurence of cardiovascular events | From date of enrollment up to 36 months
  Non-fatal cardiovascular events
The Incidence of new diabetic complications | From date of enrollment up to 36 months
  The onset of new micro and macrovascular complications of diabetes will be recorded
Change in soluble suppression of tumorigenesis-2 levels | From date of enrollment up to 36 months
  The levels of soluble suppression of tumorigenesis-2 will be analyzed.
Change in N-terminal pro-B-natriuretic peptide levels | From date of enrollment up to 36 months
  The levels of N-terminal pro-B-natriuretic peptide will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Tortato, MD, Principal Investigator — IRCCS INRCA, Ancona, Italy
Locations (1):
- IRCCS INRCA Hospital, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No